CLINICAL TRIAL: NCT03158779
Title: Phase II Trial Evaluating Stereotactic Body Radiation Therapy (SBRT) After Induction Chemotherapy for Patients With Locally Advanced Unresectable Pancreatic Cancer
Brief Title: Evaluation of SBRT for Patients With Locally Advanced Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1736
Record Dates: First submitted 2017-05-04; First posted 2017-05-18 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT and chemotherapy (Experimental): Participants received 4 months of FOLFIRINOX or Gemcitabine-Abraxane before SBRT was administered. A 3-weeks break from chemotherapy and restaging with thorax-abdominal CT scan to confirm the absence of distant metastases was required before SBRT delivery.
  Before SBRT simulation, patients may will have implanted fiducial into the pancreatic tumor.
  The SBRT schedule will be [6 x 9 Gy = 54 Gy] delivered in consecutive days.
  Interventions: Combination Product: SBRT and chemotherapy

INTERVENTIONS:
Combination Product: SBRT and chemotherapy — Patients affected by locally unresectable pancreatic cancer receive integrated treatment of FOLFIRINOX or Gemcitabine-Abraxane and a Stereotactic Body Radiation Therapy with a total dose of 54 Gy in 6 fractions of 9 Gy /fractions.

SUMMARY:
The aim of this phase II study is to assess the efficacy and safety of sequentially integrated treatment of FOLFIRINOX or Gemcitabine-Abraxane and SBRT in patients with unresectable pancreatic cancer.

DETAILED DESCRIPTION:
The aim of this prospective mono-institutional phase II study is to assess the efficacy and safety of sequentially integrated treatment of FOLFIRINOX or Gemcitabine-Abraxane and SBRT with a total dose of 54 Gy in 6 fractions of 9 Gy /fractions in patients with locally unresectable pancreatic cancer.

Primary endpoint is to evaluate overall survival (OS); the overall survival time will be calculated from the start of chemotherapy to death. Secondary end points are to evaluate acute and late toxicities, freedom from local progression (FFLP) and progression free-survival (PFS). Acute and late toxicities will be scored according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Local progression will be defined according to RECIST criteria. Time to toxicity and time to local or distant progression will be defined from the start of chemotherapy.

Technical success will be defined as the ability to implant at least 2 fiducials in the tumor area. Migration will be defined as a change in inter-fiducial distance. Clinical success will be defined as the ability to guide the application of SBRT by using the fiducials. Any adverse event will be recorded (acute pancreatitis, clinically relevant upper GI bleeding requiring blood transfusion, abscesses in the area of the fiducials, sepsis).

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or radiologically (CT scan and/or MRI scan and/or FDG-PET) proven unresectable locally advanced pancreatic cancer, discussed multidisciplinary by tumor board.
* Eighteen years of age or older,
* Minimum Karnofsky Performance Status of 70.
* Lesions cannot exceed 5 cm in maximum diameter.
* Absence of lymph-nodal metastases
* Patients received 4-6 months of FOLFIRINOX or Gemcitabine-Abraxane before SBRT was administered.
* Baseline total body CT scan performed no more than 2 months before treatment.
* Placing fiducial markers through endoscopes is permitted (EUS-guided fiducials placement before the treatment).
* Acceptable organ and bone marrow function.
* Ability to maintain the set-up position during RT.
* All patients give informed consent and sign a study-specific informed consent form.

Exclusion Criteria:

* Metastatic disease
* Prior abdominal radiotherapy
* Other malignancies diagnosed within 5 years
* Gastric or duodenal obstruction.
* Concurrent chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Evaluation of SBRT after induction CT with FOLFIRINOX or Gemcitabine-Abraxane in terms of overall survival time that will be calculated from the start of chemotherapy to death.

SECONDARY OUTCOMES:
Incidence of acute toxicities | 2 years
  Evaluation of early post treatment complications according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Incidence of late toxicities | 4 years
  Evaluation of late post treatment complications according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Freedom from local progression in treated patients | 2 years
  Evaluation of proportion of patients free from local progression according to RECIST criteria
Progression free-survival of treated patients | 2 years
  Evaluation of proportions of patients alive and free form progression according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marta Scorsetti, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No